CLINICAL TRIAL: NCT05197790
Title: A Single Center Study on the Functionality of the Pulse Oximeter and Accelerometer Portions of a Novel Wearable Device
Brief Title: Functionality of the Pulse Oximeter and Accelerometer Portions of a Novel Wearable Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 849910
Record Dates: First submitted 2021-12-10; First posted 2022-01-20 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Hypoxic Events

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Assess device prototype functionality (Other): Everyone will be in the same arm
  Interventions: Device: FDA approved pulse oximeter and DOVE device prototype

INTERVENTIONS:
Device: FDA approved pulse oximeter and DOVE device prototype — The objective is to assess reasonable detection of hypoxic episodes

SUMMARY:
The purpose of this study is to asses the function of an oxygen sensor and the movement sensor in a novel device prototype.

DETAILED DESCRIPTION:
After informing the patient about the study and the potential risk. The patient is asked to wear a prototype of a novel device to sense oxygen levels and movement for the duration of the visit. The day of the enrolment is when the visit will be completed. The patient is required to complete an overnight sleep test (no more than 15 hrs) with the prototype device worn on their index finger and wrist.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* 21 years of age or older
* Suspected to suffer from hypoxic events
* Able to provide informed consent

Exclusion Criteria:

* Pregnant

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2024-12-21 (Actual); Study Completion 2024-12-28 (Actual)

PRIMARY OUTCOMES:
Comparing Dove device against FDA approved SpO2 sensor | 15 hours
  Dove device will be analyzed against FDA approved SpO2 and Skin tone will be incorporated as a factor of SpO2 function to ensure the device can be reasonably detect hypoxia.

SECONDARY OUTCOMES:
Questionnaire about comfort of device | 15-20 minutes depending on the patients questions.
  Participant will be surveyed for their subjective comfort wearing the DOVE prototype device. The questionnaire will ensure topics such as compliance and comfort or any issues and experiences the subject had with the prototype device.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States